CLINICAL TRIAL: NCT04460170
Title: COVID-19 Follow up Intensive Care Studies
Acronym: COFICS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hanze University of Applied Sciences Groningen (Other)
Responsible Party: Principal Investigator, Willem Dieperink, PhD, University Medical Center Groningen
Other Study IDs: COFICS201800422
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Quality of Life; COVID-19
Keywords: Critical Care; Family Members; Patients; Follow-Up Studies; Quality of Life; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the SARS-CoV-2 infection is relatively new, the long term attributable burden related to COVID19 has not been investigated yet. To date, in patients with COVID-19 and their family members, there is little information on the functional status, cognitive ability, pattern of return to work, and health related quality of life after the ICU admission.

This study aims to describe the psychological wellbeing, physical - and social functioning of COVID-19 ICU survivors and their family members up to 12 months following ICU discharge.

DETAILED DESCRIPTION:
Study design The COVID-19 Follow up Intensive Care Study (COFICS) is a single center, prospective cohort study performed at a University Medical Center in The Netherlands.

Study population The study population consists of all admitted critically ill COVID-19 patients with a > 48 hours ICU admission at the ICU of a University Medical Center and a family member of the patient. Family members in this study can be partners, other family members, or friends who are identified by the patient as important.

Sample size All consecutive patients admitted to the ICU of the University Hospital for respiratory distress due to COVID-19 between March 19th 2020 and September 30th 2020 will be enrolled. With consent of the patient, family member(s) of participating patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Ability to speak and write Dutch
* Ability to conduct a telephone call
* Diagnosed with COVID-19 infection (only in patients)
* 48 hours ICU admission (only in patients)

Exclusion Criteria:

* Refuse to participate
* Serious language barrier
* Cognitive impairment
* Severe psychiatric disorder
* Chronic ventilator dependency (only in patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all admitted critically ill COVID-19 patients with a > 48 hours ICU admission at the ICU of a University Medical Center and a family member of the patient. Family members in this study can be partners, other family members, or friends who are identified by the patient as important.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
General Health | 3 months post ICU discharge
  MOS Short-Form General Health Survey (SF-20). The SF-20 contains 20 items and has six dimensions; physical functioning (min. score 6, max. score 12) rolefunctioning (min. score 2, max. score 4) social functioning (min. score 1, max. score 6) mental health (min. score 5, max. score 30) general health (min. score 5, max. score 25) pain (min. score 1, max score 5) All endscores will be transformed to a 100 points scale where a higher score means better functioning. Except for pain where a higher score means more pain.
  The five mental health questions will be excluded from our questionnaire because the questions are comparable with the HADS.
General Health | 6 months post ICU discharge
  MOS Short-Form General Health Survey (SF-20). The SF-20 contains 20 items and has six dimensions; physical functioning (min. score 6, max. score 12) rolefunctioning (min. score 2, max. score 4) social functioning (min. score 1, max. score 6) mental health (min. score 5, max. score 30) general health (min. score 5, max. score 25) pain (min. score 1, max score 5) All endscores will be transformed to a 100 points scale where a higher score means better functioning. Except for pain where a higher score means more pain.
  The five mental health questions will be excluded from our questionnaire because the questions are comparable with the HADS.
General Health | 12 months post ICU discharge
  MOS Short-Form General Health Survey (SF-20). The SF-20 contains 20 items and has six dimensions; physical functioning (min. score 6, max. score 12) rolefunctioning (min. score 2, max. score 4) social functioning (min. score 1, max. score 6) mental health (min. score 5, max. score 30) general health (min. score 5, max. score 25) pain (min. score 1, max score 5) All endscores will be transformed to a 100 points scale where a higher score means better functioning. Except for pain where a higher score means more pain.
  The five mental health questions will be excluded from our questionnaire because the questions are comparable with the HADS.
Anxiety and Depression | 3 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS). The HADS contains two subscale of 7 items each. Minimal score is 0, maximal score 21 for each subscale where a higher score means a higher burden.
Anxiety and Depression | 6 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS). The HADS contains two subscale of 7 items each. Minimal score is 0, maximal score 21 for each subscale where a higher score means a higher burden.
Anxiety and Depression | 12 months post ICU discharge
  Hospital Anxiety and Depression Scale (HADS). The HADS contains two subscale of 7 items each. Minimal score is 0, maximal score 21 for each subscale where a higher score means a higher burden.
Long function | 6 months post ICU discharge (only in patients)
  Spirometry test
Long function | 12 months post ICU discharge (only in patients)
  Spirometry test
Frailty | 3 months post ICU discharge (only in patients)
  Clinical Frailty Scale with a single outcome measure summarizing the overall level of fitness.
Frailty | 6 months post ICU discharge (only in patients)
  Clinical Frailty Scale with a single outcome measure summarizing the overall level of fitness.
Frailty | 12 months post ICU discharge (only in patients)
  Clinical Frailty Scale with a single outcome measure summarizing the overall level of fitness.
Family functioning | 6 months post ICU discharge
  McMaster Family Assessment Device (FAD-GF6+). The FAD-GF6+ contains 6 items (min. score 6, max. score 24) where a higher scores indicate a lower caregiver burden.
Family functioning | 12 months post ICU discharge
  McMaster Family Assessment Device (FAD-GF6+). The FAD-GF6+ contains 6 items (min. score 6, max. score 24) where a higher scores indicate a lower caregiver burden.
Effect of an ICU admission on return to work | 3 months post ICU discharge (only in family members)
  Return to work knowing; possible job loss, change of work activities and worsening employment status
Effect of an ICU admission on return to work | 6 months post ICU discharge
  Return to work knowing; possible job loss, change of work activities and worsening employment status
Effect of an ICU admission on return to work | 12 months post ICU discharge
  Return to work knowing; possible job loss, change of work activities and worsening employment status

SECONDARY OUTCOMES:
age | 24 hours (patient) / 3 months post ICU discharge (family member)
  age (years)
Gender | 24 hours (patient) / 3 months post ICU discharge (family member)
  Gender (male/female)
Social status | 3 months post ICU discharge
  Social status (married/living together/ single)
APACHE IV | 24 hours (only in patients)
  Acute Physiology And Chronic Health Evaluation (APACHE IV). It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): based on several measurements; higher scores correspond to more severe disease and a higher risk of death
Comorbidity | 3 months post ICU discharge (only in patients)
  Comorbidity ( free text)
Body mass index | 3 months post ICU discharge (only in patients)
  Body mass index (kg/m2)
ICU stay | hospital discharge, an average of 4 weeks (only in patients)
  ICU stay (days)
Mechanical ventilation | hospital discharge, an average of 4 weeks (only in patients)
  Mechanical ventilation (days)
Delerium | hospital discharge, an average of 4 weeks (only in patients)
  Delerium (no / yes --> CAM-ICU / DOS score)
Hospital stay | hospital discharge, an average of 4 weeks (only in patients)
  Hospital stay (days)
Discharge locationn | hospital discharge, an average of 4 weeks (only in patients)
  Discharge location (home, other hospital, nursing home, revelidation center)
Mortality | 3 months post ICU discharge (only in patients)
  Mortality (no / yes --> date)
Mortality | 6 months post ICU discharge (only in patients)
  Mortality (no / yes --> date)
Mortality | 12 months post ICU discharge (only in patients)
  Mortality (no / yes --> date)
Relationship with the patient | 3 months post ICU discharge (only in family members)
  Relationship with the patient (Partner, sibling, child, other)
Educational level | 3 months post ICU discharge
  Educational level (low, middle, high)
Readmission | 3 months post ICU discharge (only in patients)
  Readmission (no / yes --> free text)
Health care consumption | 3 months post ICU discharge
  Health care consumption (general practicionar, home care, physiotherapist, lung specialist, psychologist, onther (free text))
Health care consumption | 6 months post ICU discharge
  Health care consumption (general practicionar, home care, physiotherapist, lung specialist, psychologist, onther (free text))
Health care consumption | 12 months post ICU discharge
  Health care consumption (general practicionar, home care, physiotherapist, lung specialist, psychologist, onther (free text))
Weight | 3 months post ICU discharge
  Weight (kg)
Weight | 6 months post ICU discharge
  Weight (kg)
Weight | 12 months post ICU discharge
  Weight (kg)
Hypertensive | 3 months post ICU discharge
  Hypertensive (RR)
Hypertensive | 6 months post ICU discharge
  Hypertensive (RR)
Hypertensive | 12 months post ICU discharge
  Hypertensive (RR)
Thrombosis | 3 months post ICU discharge
  Thrombosis (no / yes --> anticoagulant, DVT or PE)
Thrombosis | 6 months post ICU discharge
  Thrombosis (no / yes --> anticoagulant, DVT or PE)
Thrombosis | 12 months post ICU discharge
  Thrombosis (no / yes --> anticoagulant, DVT or PE)
Diabetes | 3 months post ICU discharge
  Diabetes (no /yes --> current insulin level, metformin/ insulin use)
Diabetes | 6 months post ICU discharge
  Diabetes (no /yes --> current insulin level, metformin/ insulin use)
Diabetes | 12 months post ICU discharge
  Diabetes (no /yes --> current insulin level, metformin/ insulin use)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands